CLINICAL TRIAL: NCT03978481
Title: Effect of Helicobacter Pylori Eradication After Subtotal Gastrectomy on Survival Rate of Gastric Cancer Patients: Retrospective Study
Status: Completed | Type: Observational
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Nayoung Kim, Professor, Seoul National University Bundang Hospital
Other Study IDs: B-1902-523-107
Record Dates: First submitted 2019-06-02; First posted 2019-06-07 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2021-03

CONDITIONS: Gastric Cancer
Keywords: Gastric cancer; Helicobacter pylori; Subtotal gastrectomy; Overall survival; Metachronous cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Combined Modality Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Eradicated group: Gastric cancer patients received subtotal gastrectomy, with Helicobacter pylori eradication
  Interventions: Combination Product: Helicobacter pylori eradication (combination therapy)
- Negative group: Gastric cancer patients received subtotal gastrectomy, without Helicobacter pylori eradication or Helicobacter pylori negative

INTERVENTIONS:
Combination Product: Helicobacter pylori eradication (combination therapy) — Antibiotic eradication therapy (triple or quadriple regimen)
  Groups: Eradicated group

SUMMARY:
In this study, we will observe the long-term survival rate, overall mortality rate, gastric cancer specific mortality rate, and the incidence rate of metachronous cancer in patients who received subtotal gastrectomy, with or without Helicobacter pylori eradication.

DETAILED DESCRIPTION:
In this study, we will observe the long-term survival rate, overall mortality rate, gastric cancer specific mortality rate, and the incidence rate of metachronous cancer in patients who received subtotal gastrectomy, with or without Helicobacter pylori eradication. In addition, we will analyze the correlation between the incidence and survival rate of this type of stomach cancer by comparing smoking, gastric cancer direct family history, disease stage (TNM staging), the histologic type of stomach cancer (intestinal, diffuse, mixed), and the surgical method (Billoth I, Billoth II) as well as the infection and eradication status of H. pylori.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with gastric cancer and received surgery (partial, distal, subtotal gastrectomy), and tested Helicobacter pylori status

Exclusion Criteria:

* Patients with other severe diseases (other primary cancer, severe cardiovascular, cerebral, renal, hepatic diseases)
* Patients received palliative treatment

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with gastric cancer and received surgery (partial, distal, subtotal gastrectomy), and tested Helicobacter pylori status in Seoul National University Bundang Hospital, from 2003 to 2018
Sampling Method: Non-Probability Sample
Enrollment: 3700 (Actual)
Dates: Start 2019-01-30 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Overall survival | From date of initial curative surgery for gastric cancer, until the date of death from any cause, up to 60 months

SECONDARY OUTCOMES:
Gastric cancer-specific (disease-free) survival | From date of initial curative surgery for gastric cancer, until the date of diagnosis of gastric cancer recurrence or the date of death, whichever comes first, up to 60 months
  Survival period without cancer recurrence or newly developed stomach cancer diagnosis
Metachronous cancer (remnant stomach cancer) | Up to 60 months
  The number of patients who were diagnosed with new carcinoma on the remnant stomach, over follow-up period of up to 60 months, in eradication group and non-eradication group

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: Undecided